CLINICAL TRIAL: NCT04641559
Title: Personalized Nutrition Advice Based on Metabolic Profiling and Behaviour Assessment for Optimizing Dietary Habits and Metabolic Status. Single Blind, Parallel, Randomized, Controled Intervention Trial (EUT_PREVENTOMICS)
Brief Title: Personalized Nutrition Advice for Optimizing Dietary Habits and Metabolic Status
Acronym: PREVENTOMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other); Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EUT_PREVENTOMICS
Record Dates: First submitted 2020-11-02; First posted 2020-11-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Personalized Nutrition; Health Status; Dietary Habits
Keywords: Metabolic status; gut microbiota; Behavioural intervention; Mediterranean diet; Retailer website; Preventomics; Digital environment
MeSH Terms: conditions — Feeding Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized nutrition group (Experimental): Intervention group that will receive personalized nutrition advice through the ALDI's catalogue during four months.
  Interventions: Other: Personalized nutrition group
- Personalized Plan group (Experimental): Intervention group that will receive personalized nutrition advice through the ALDI's catalogue and behavioural change program during four months.
  Interventions: Other: Personalized Plan group
- Control group (Placebo Comparator): General recommendations but not personalization nor behavioural change advice will be implemented during four months.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Personalized nutrition group — A digital environment which combines biological information, personal habits and preference to provide nutritional recommendations. This digital environment is composed by the follow softwares:1. The recommender system: software that combine the behavioral and biological information about the volunteer and generates personalized nutritional recommendations; 2. The ALDI microsite: A microsite that retrieves the personalized recommendations for the volunteer from the recommender system. The ALDI microsite matches food categories with products of the ALDI catalogue. As a result, the volunteer receives a list of products classified under different food categories that are recommended for him/her. Next to each food category, the number of servings recommended (weekly or daily) is also shown.
  The ALDI microsite is a tool only to elaborate a shopping list through personalized recommendations. Therefore, volunteers can choose to buy their food shopping list at wherever store other from ALDI.
  Arms: Personalized nutrition group
Other: Personalized Plan group — Participants will use the same software described in for the Personalized nutrition group together with a behavioral change program designed to increase the adherence to the recommendations provided by the ALDI microsite by promoting a proper attitude by means of a series of personalized, goal-orientated, friendly, achievable actions delivered periodically to the volunteer. The behavioral change program will be fed with the results of behavior questionnaires. The personalized messages will be delivered through the ALDI microsite. These personalized messages will be available only for those subjects engaged in the Personalized Plan group.
  Arms: Personalized Plan group
Other: Control group — The participants in the control group will not have personalized recommendations. These participants will have access to a restricted version of the ALDI microsite where the list of recommended products correspond to categories that are general recommendations according to Mediterranean diet.
  Arms: Control group

SUMMARY:
The alteration maintained over time of some metabolic processes, such as oxidative stress, low-grade inflammation, carbohydrate and lipid metabolism, and of the intestinal microbiota activity, can induce some chronic diseases with high prevalence in society, such as obesity, cardiovascular disease or diabetes. These metabolic alterations can be modulated through nutrition and eating habits. Thus nutritional interventions are currently considered as a main tool for disease prevention.

The need to adapt nutritional interventions to the particular needs of each person in order to improve the health status of all individuals is becoming more and more evident, through precision nutrition. On the other hand, for nutritional interventions to be carried out over long periods of time and to achieve sustainable long-term changes in lifestyle, new forms of behavioral counseling are necessary to facilitate the follow-up of nutritional interventions.

PREVENTOMICS is a European project that arose to develop a personalized nutrition system, the PREVENTOMICS system. This system is based on the classification of the users of the system according to the state of their own metabolic processes, their genotype, their dietary habits and preferences, levels of physical activity, purchase preference and possible allergies, in order to provide a personalized nutrition adapted to the needs of each user.

The PREVENTOMICS system is presented through a digital environment via computer, with a list of products provided by the ALDI supermarket to prepare the shopping list, without having to buy the products from the ALDI supermarket.

DETAILED DESCRIPTION:
Nowadays, diet is recognized as one of the most important factors in the development of non-communicable diseases. Therefore, nutrition and dietary habits stand out as an invaluable tool for preventing diseases. Among these dietary habits, Mediterranean diet is now recognized as one of the best models of food patterns providing protection against chronic diseases and with beneficial effects on quality of life.

During the last years, expectation on precision nutrition beyond personalized diet has been increasing due to the possibility of adapting diet to the actual needs of the person, optimizing the function of the organism. Currently, diet precision in the context of general population is mainly addressed to heterogeneous groups of population, depending on variables such as age, gender or physical state among others. Beyond this approach, a more accurate personalization strategy is based on adapting some components of the diet to the genetic profile of the subject while considering a limited number of phenotypical traits.

Some authors have proposed that a wide array of chronic non-communicable diseases of high prevalence in our society have a multifactorial origin, being the result of a sustained dysregulation of some physiological processes, such as metabolic stress, oxidative stress, chronic systemic low-grade inflammation or psychological stress among others. Since most of these processes can be modulated by diet, optimizing them by means of nutritional interventions could represent an invaluable approach for preventing diseases. Nevertheless, a complete characterization of these physiological processes is needed in order to know their real state in individuals and be able to deliver an adequate intervention for their restoration when required. Currently, -omics technologies provide the necessary tools for accurate assessing the state of these physiological processes.

In this context, PREVENTOMICS project financed by the European Research and Innovation programme H2020 (Call H2020-SFS-2018-2020; DT-SFS-14-2018; Project title : Empowering consumers to PREVENT diet-related diseases through OMICS sciences) and with a consortium of different companies and public entities, including EURECAT, aims to assess the most relevant metabolic processes which dysregulation leads to the onset of disease and to integrate individual's metabolic signature with genetic, biological, nutritional and psychological aspects through Information and communication Technologies (ICTs) to deliver preventive personalized nutrition tools in order to correct early deviations.

The main concept behind the PREVENTOMICS project is to provide personalized recommendations based on a multi-level classification after clustering the different users according to their dietary habits and preferences, their levels of physical activity, shopping preferences, possible allergies and phenotypic (i.e. metabolomics and proteomics-based multivariate approach) and genotype characterization.

To achieve the main objective, the PREVENTOMICs project consortium has developed a personalized nutrition strategy based on a recommender system in order to provide personalized nutrition tailored to the actual status of the subject.

To do that, the physiological processes considered in PREVENTOMICS have been selected according to their relevance with health and disease, to nutritional status and, therefore, their ability for being modulated by nutritional interventions.

These processes are:1) oxidative stress; 2) systemic inflammation; 3) carbohydrate metabolism; 4) lipid metabolism; 5) microbiota status through the measurement of microbiota generated metabolites.

In order to define the status of these physiological process, classically accepted biomarkers already used in clinical assessment and intervention studies will be determined, including blood triglycerides, cholesterol, C-reactive protein, glucose or urine isoprostanes among others. Moreover, the recommender system developed in PREVENTOMICS combines these measurements with other biomarkers that have been sufficiently well characterized as surrogates for studying specific metabolic processes.

With the above information, the PREVENTOMICS recommender system also integrates a panel of single nucleotide polymorphisms (SNPs).

Besides, behavioural research shows clearly that the provision of knowledge and advice as a means to help people make changes in their lifestyles does not necessarily result in the desired behavioural change. Therefore, in order to achieve sustainable long-term lifestyle changes, people need to be prompted to behave in new ways that do not rely on their willpower or conscious thinking.

Therefore, the recommender system will anonymously collect data on analyzed biomarkers, habits, mental wellbeing levels, cognitive health, social inclusion and behaviours and will translate this using behavioural change algorithms along with digital delivery into a series of personalised, goal-orientated, friendly, and achievable actions proposed to the user.

Thus, to achieve PREVENTOMICS project objectives, a consortium of 19 partners was created including:

1. 4 small medium-sized enterprises (Alimentomica, Carinsa, Do Something Different and Practico);
2. 9 research performing institutions (Eurecat, University of Parma, University of Southampton-Southampton General Hospital, Institute of Communication and Computer Systems, Maastrich University, Wageningen University, Leitat, Jagiellonian University Medical College);
3. 3 companies with exploitation interests (SimpleFeast, Meteda and Aldi)
4. A consumer association OCU;
5. A standardization body, UNE;
6. Osteoarthritis Foundation International - OAFI.

The main outcome of the PREVENTOMICS project has been a novel recommender system that can be used in a wide array of applications or business models. Within the PREVENTOMIC project, three different applications of the system are evaluated:

1. Personalization of weekly menus delivered at home (catering).
2. Adaptation of professional tools for nutritionists and dieticians (advanced tools for health professionals).
3. Personalized shopping experience in supermarket (retailers).

In PREVENTOMICS project, the UTNS of Eurecat in Reus is focused in personalized shopping experience together with ALDI supermarkets and will conduct the study with clinically healthy adults and using a dedicated ALDI microwebsite to assess application number 3.

The ALDI microsite uses the personalized recommendations generated by the recommender system to provide each user the most appropriate diet-based nutritional and behavioural changes recommendations according to the individual's needs, lifestyle and preferences and personalizing the shopping experience in ALDI's online supermarket.

Importantly, despite the proposed use of such workflow might be demonstration of personalized online shopping, the pilot carried out in Reus does not support trading. Therefore, users will use the ALDI microsite to generate a shopping list navigating through a personalized ALDI catalog, but they are free to shop at any retailer other than ALDI.

The improvement in dietary habits will be based on the Mediterranean diet adherence as a reference, as this diet is recognized as one gold standard.

The hypothesis of the present study is that empowering consumers with tools that adapt nutrition recommendations to individual's metabolic state, lifestyle and food preferences through the utilization of the recommender system developed in PREVENTOMICS, with or without the application of behavioral change programs, will promote favorable and sustained changes in personal dietary behavior and food choices at the supermarket, promoting Mediterranean diet and beneficial effects on the health status of individuals.

The main objective of the present study is to assess the soundness of the personalized nutrition advice generated by the recommender system and its combination with a behavioral change intervention, to improve dietary habits of individuals compared to standard and generic nutritional advice, measured through adherence to the Mediterranean diet and delivered through a retailer website (ALDI microsite).

The secondary objectives are to evaluate the effects of using the personalized nutrition advice provided by PREVENTOMICS through a retailer website on:

* Anthropometric measurements.
* Blood pressure.
* Metabolic profile.

After the selection visit (V0), on the first visit (V1), the 180 participants will provide urine, stool and saliva samples and will fill different questionnaires (quality of life, behavior, frequency of food consumption and physical activity) with the help of nutritionists. Additionally, participants will be randomly divided into three groups of 60 participants as they receive: 1) personalized nutritional advice; 2) personalized nutritional and behavior change advice; or 3) general non-personalized nutritional advice. With the samples provided in the first visit, a complete analysis of the metabolic and genetic status of each participant will be carried out, which will be used for, approximately after a month, the participant begins to use the digital environment to generate their shopping list. Users will follow the nutritional advice that corresponds to them according to the assigned group and through the PREVENTOMICS system for 4 months. After 4 months, participants will make the last study visit (V2) where they will repeat the same process described for the first visit to assess the effects of the intervention.

During the study, 3 visits will be carried out:

* One selection visit (V0; week 1) to check inclusion / exclusion criteria in the study and provide the necessary material for collecting stool and urine samples, as well as a three-day dietary record.
* A visit start of the study (V1; week 2) in which the participant will bring the biological samples, will fill the questionnaires and three-day dietary record, will have blood drawn and obtain a saliva sample, and will be included in one of the three study groups.
* A visit of completion of the study (V2; week 25), in which the participant will bring the biological samples, will have blood drawn and will fill out the questionnaires and three-day dietary record.

Monthly, except for the last month of the study, the participant will be followed up by phone call. In the last one, there will be a face-to-face follow-up visit to give the volunteers the materials for collecting biological samples and the three-day dietary record for the V2 visit. In addition, the participants will have personalized support by phone and via email for any questions or problems that may arise during the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Signed informed consent.
* To have internet access.

Exclusion Criteria:

* Diabetes (or glucose ≥ 126 mg/dL or pharmacological treatment).
* Hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg or pharmacological treatment).
* Dyslipidaemia (cLDL ≥4.9 mmol/L and/or triglycerides ≥4.5 mmol/L (≥400 mg/dL) and/or cHDL <40 mg/dL (1.03 mmol/L) in men and <50 mg/dL (1.29 mmol/L) in women) or with pharmacological treatment.
* Use of prescribed medicine to control acute or chronic inflammation.
* Anaemia (haemoglobin ≤13 g/dL in men and ≤12 g/dL in women)
* BMI (in kg/m2) <18.5 or >35.
* Being pregnant or planning to become pregnant within the study period.
* Be in breastfeeding period.
* Current smokers.
* Participate in or have participate in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
* Present some chronic gastrointestinal disease.
* Present some chronic disease with clinical manifestation, like coronary heart diseases, cardiovascular disease, coeliac disease, Crohn's disease and chronic kidney disease (or serum creatinine ≥1.7 mg/dL for men and ≥1.5 mg/dL for women).
* Following a prescribed diet for any reason, including weight loss, in the last 3 months.
* Following a pharmacological treatment for weight loss or intake of food supplements or medications that could affect body weight.
* Having allergies or food intolerances.
* No or limited access to the Internet.
* Consumption of more than 14 drinks of alcoholic beverages per week.
* Mediterranean Diet Adherence Score (MEDAS) > 8 of 14 points, which is a food pattern already highly concordant with the Mediterranean Diet.
* Being unable to follow the study guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to Mediterranean diet. | At weeks 2 and 25.
  Adherence to Mediterranean diet measured through the MEditerranean Diet Adherence Screener (MEDAS). The questionnaire consists of 14 questions about eating habits, the frequency of consumption of typical foods of the Mediterranean diet or the consumption of foods not recommended in this diet. Each question is screened with 0 (non-compliant) or 1 (compliant) and the total score range from 0 to 14, so a score of 14 points mean maximum adherence.

SECONDARY OUTCOMES:
Change in body weight. | At weeks 2 and 25
  Body weight measured by TANITA SC330.
Height. | At weeks 2
  Height measured by standardized methods.
Change in BMI | At weeks 2 and 25
  Weight and Height will be combined to report BMI in kg/m^2.
Change in waist circumference. | At weeks 2 and 25
  Waist circumference using a measuring tape.
Change in blood pressure (in mmHg). | At weeks 2 and 25
  Systolic and systolic blood pressure will be measured twice after 2-5 minutes of patient respite, seated, with one-minute interval in between, using an automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Change in urinalysis. | At weeks 2 and 25
  Urine urinalysis will be measured by standardized methods in Cobas Mira Plus autoanalyzer .(Roche Diagnostics Systems, Madrid, Spain).
Change in blood cell count. | At weeks 2 and 25
  Blood cell count will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum creatinine levels. | At weeks 2 and 25
  Serum creatinine levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum urea levels. | At weeks 2 and 25
  Serum urea levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum uric acid levels. | At weeks 2 and 25
  Serum uric acid levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum bilirubin levels. | At weeks 2 and 25
  Serum bilirubin levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum ions levels. | At weeks 2 and 25
  Serum ions levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum proteins levels. | At weeks 2 and 25
  Serum proteins levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum aspartate aminotransferase levels. | At weeks 2 and 25
  Serum aspartate aminotransferase levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in serum alanine aminotransferase levels. | At weeks 2 and 25
  Serum alanine aminotransferase levels will be measured by standardized methods in Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain).
Change in plasma IL-6 levels. | At weeks 2 and 25
  Plasma IL-6 levels will be measured by human ELISA kits.
Change in plasma TNFα levels. | At weeks 2 and 25
  Plasma TNFα levels will be measured by human ELISA kits.
Change in plasma MCP-1 levels. | At weeks 2 and 25
  Plasma MCP-1 levels will be measured by human ELISA kits.
Change in plasma IL-8 levels. | At weeks 2 and 25
  Plasma IL-8 levels will be measured by human ELISA kits.
Change in plasma soluble ICAM1 levels. | At weeks 2 and 25
  Plasma soluble ICAM1 levels will be measured by human ELISA kits.
Change in plasma soluble CD14 levels. | At weeks 2 and 25
  Plasma soluble CD14 levels will be measured by human ELISA kits.
Change in urine N-acetylglycoproteins levels. | At weeks 2 and 25
  Urine N-acetylglycoproteins levels will be measured using proton nuclear magnetic resonance.
Change in urine fucose levels. | At weeks 2 and 25
  Urine fucose levels will be measured using proton nuclear magnetic resonance.
Change in serum total PUFAs levels. | At weeks 2 and 25
  Serum total PUFAs levels will be measured using proton nuclear magnetic resonance.
Change in serum ARA and EPA levels. | At weeks 2 and 25
  Serum ARA and EPA levels will be measured using proton nuclear magnetic resonance.
Change in serum DHA levels. | At weeks 2 and 25
  Serum DHA levels will be measured using proton nuclear magnetic resonance.
Change in serum linoleic acid levels. | At weeks 2 and 25
  Serum linoleic acid levels will be measured using proton nuclear magnetic resonance.
Change in plasma lysophosphatidylcholine levels. | At weeks 2 and 25
  Plasma lysophosphatidylcholine levels will be measured using proton nuclear magnetic resonance.
Change in serum acetate levels. | At weeks 2 and 25
  Serum acetate levels will be measured using proton nuclear magnetic resonance.
Change in urine acetate levels. | At weeks 2 and 25
  Urine acetate levels will be measured using proton nuclear magnetic resonance.
Change in serum lactate levels. | At weeks 2 and 25
  Serum lactate levels will be measured using proton nuclear magnetic resonance.
Change in urine lactate levels. | At weeks 2 and 25
  Urine lactate levels will be measured using proton nuclear magnetic resonance.
Change in urine TMAO levels. | At weeks 2 and 25
  Urine TMAO levels will be measured using proton nuclear magnetic resonance.
Change in urine TMA levels. | At weeks 2 and 25
  Urine TMA levels will be measured using proton nuclear magnetic resonance.
Change in urine DMA levels. | At weeks 2 and 25
  Urine TMA levels will be measured using proton nuclear magnetic resonance.
Change in plasma LPS levels. | At weeks 2 and 25
  Plasma LPS levels will be measured using gas chromatography mass spectrometry.
Change in plasma glucose levels | At weeks 2 and 25
  Plasma glucose levels will be measured by enzymatic methods.
Change in plasma insulin levels | At weeks 2 and 25
  Plasma insulin levels will be measured by human ELISA kits.
Change in plasma leptin levels | At weeks 2 and 25
  Plasma leptin levels will be measured by human ELISA kits.
Change in plasma adiponectin levels | At weeks 2 and 25
  Plasma adiponectin levels will be measured by human ELISA kits.
Change in urine α-hydroxybutyrate levels | At weeks 2 and 25
  Urine α-hydroxybutyrate levels will be measured using proton nuclear magnetic resonance.
Change in urine α-ketoglutarate levels | At weeks 2 and 25
  Urine α-ketoglutarate levels will be measured using proton nuclear magnetic resonance.
Change in urine fumarate levels | At weeks 2 and 25
  Urine fumarate levels will be measured using proton nuclear magnetic resonance.
Change in urine succinate levels | At weeks 2 and 25
  Urine succinate levels will be measured using proton nuclear magnetic resonance.
Change in urine malate levels | At weeks 2 and 25
  Urine malate levels will be measured using proton nuclear magnetic resonance.
Change in plasma acylcarnitine profile levels | At weeks 2 and 25
  Plasma acylcarnitine profile levels will be measured by liquid chromatography mass spectrometry.
Change in HOMA-IR levels | At weeks 2 and 25
  HOMA-IR will be measured based on fasting blood levels of glucose an insulin.
Change in leptin to adiponectin ratio | At weeks 2 and 25
  Leptin to adiponectin ratio will be calculated using blood levels of leptin ad adiponectin.
Change in plasma total cholesterol levels | At weeks 2 and 25
  Plasma total cholesterol levels will be measured by enzymatic methods.
Change in plasma HDL-cholesterol levels | At weeks 2 and 25
  Plasma HDL-cholesterol levels will be measured by enzymatic methods.
Change in plasma non-HDL-cholesterol levels | At weeks 2 and 25
  Plasma non-HDL-cholesterol levels will be measured by enzymatic methods.
Change in plasma triglycerides levels | At weeks 2 and 25
  Plasma triglycerides levels will be measured by enzymatic methods.
Change in plasma LDL-cholesterol levels | At weeks 2 and 25
  Plasma LDL-cholesterol levels will be measured using the Friedwald formula.
Change in the atherogenic index of plasma | At weeks 2 and 25
  The atherogenic index of plasma will be calculated as log(TG/HDL-cholesterol).
Change in serum total MUFAs levels | At weeks 2 and 25
  Serum total MUFAs levels will be measured using proton nuclear magnetic resonance.
Change in serum oleic acid levels | At weeks 2 and 25
  Serum oleic acid levels will be measured using proton nuclear magnetic resonance.
Change in plasma total lysophosphatidylcholine levels | At weeks 2 and 25
  Plasma total lysophosphatidylcholine levels will be measured using proton nuclear magnetic resonance.
Change in urine 8-hydroxy-2'-deoxyguanosine levels | At weeks 2 and 25
  Urine 8-hydroxy-2'-deoxyguanosine levels will be measured by human ELISA kits.
Change in urine 8-iso-prostaglandin F2α levels | At weeks 2 and 25
  Urine 8-iso-prostaglandin F2α levels will be measured by human ELISA kits.
Change in plasma 3-Nitrotyrosine levels | At weeks 2 and 25
  Plasma 3-Nitrotyrosine levels will be measured by human ELISA kits.
Change in urine Pseudouridine levels | At weeks 2 and 25
  Urine Pseudouridine levels will be measured using proton nuclear magnetic resonance.
Metabolomics for consumption biomarkers | At weeks 2 and 25
  The main biomarkers of food consumption will be measured using High Resolution Liquid chromatography- tandem Mass Spectrometry (HR-LC-MS/MS) in urine.
Genotyping analysis | At week 2
  The main Single Nucleotide Polymorphisms (SNPs) related to nutrition associated disorders will be measured using oral smear and by Open Array Technology.
Change in nutrition habits | At weeks 2 and 25
  Nutritional habits and daily intake will be measured using the servings per day, week or month of the different food groups that make up the Preventomics food frequency questionnaire, an adapted food questionnaire from The European Prospective Investigation into Cancer and Nutrition (EPIC) study.
Change in physical activity | At weeks 2 and 25
  Physical activity will be evaluated through the International Physical Activity Questionnaire (IPAQ)-short for physical activity questionnaire. The questionnaire asks about three specific types of activity (walking, moderate-intensity activities and vigorous intensity activities) in the set domains leisure time, domestic and gardening (yard) activities, work-related and transport-related activities. Frequency and duration are collected separately for each specific type of activity. Both, categorical and continuous indicators will be measured.
Change in satisfaction with weight-management diets. | At weeks 2 and 25
  Quality of life will be estimated through Diet Satisfaction questionnaire (DSat-28). The questionnaire consists of 28 questions with a five point level scale with higher scores indicating greater satisfaction.
Change in person's perceptions in life related to mobility, self-care, usual activities, paint/discomfort and anxiety/depression. | At weeks 2 and 25
  Quality of life will be estimated through Euro Qol 5 Dimension (EQ-5D) questionnaire. The questionnaire consist of 28 questions with a five point scale with1 indicating the best health status and 5 indicating the worst health status, plus a visual analog score to report the perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Change in person's global perception in life related to being overweight and trying to lose weight. | At weeks 2 and 25
  Quality of life will be estimated through Obesity and Weight-Loss Quality of Life instrument (OWLQOL). The questionnaire consists of 17 statements with a six point scale, with 1 indicating the best quality of life and 6 indicating the worst quality of life.
Change in hip circumference | At weeks 2 and 25
  Hip circumference will be measured using a measuring tape
Change in body composition | At weeks 2 and 25
  Body fat mass and body lean mass (in € and in kg) will be measured using Tanita Body Composition Analyzer.
Change in dietary intake | At weeks 2 and 25
  Dietary intake will be measured using 3-day dietary record.

CONTACTS AND LOCATIONS:
Overall Officials: Josep M Del Bas, PhD, Principal Investigator — UTNS (Eurecat_Reus); Josep M Del Bas, PhD, Study Director — UTNS (Eurecat_Reus)
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing plans for the current study are unknown and will be made available at a later date

REFERENCES:
- [Derived] Calderon-Perez L, Escote X, Companys J, Alcaide-Hidalgo JM, Bosch M, Rabassa M, Crescenti A, Valls RM, Pedret A, Sola R, Marine R, Gil-Cardoso K, Rodriguez MA, Palacios H, Del Pino A, Guirro M, Canela N, Sunol D, Galofre M, Galmes S, Palou-March A, Serra F, Caimari A, Gutierrez B, Del Bas JM. A single-blinded, randomized, parallel intervention to evaluate genetics and omics-based personalized nutrition in general population via an e-commerce tool: The PREVENTOMICS e-commerce study. Am J Clin Nutr. 2024 Jul;120(1):129-144. doi: 10.1016/j.ajcnut.2024.04.004. Epub 2024 May 23. PMID 38960570
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org